CLINICAL TRIAL: NCT02438475
Title: The Safety and Efficacy of an Extravascular, Water-Soluble Sealant for Venous Access-Site Closure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Cardinal Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vascular Closure Venous Mynx
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Diagnostic Procedure; Cardiac Interventional Procedure; Femoral Access Site Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Mynx Vascular Closure System (Active Comparator): Where subjects will have venous hemostasis attempted to be achieved using the Mynx Vascular Closure system alone
  Interventions: Device: Mynx Vascular Closure System
- Manual Compression (Other): Where patients will have venous hemostasis attempted to be achieved using manual compression alone
  Interventions: Other: Manual Compression

INTERVENTIONS:
Device: Mynx Vascular Closure System — MynxGrip is being used to seal femoral vein access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F or 7F procedural sheath.
  Other Names: MynxGrip Vascular Closure Device
  Arms: Mynx Vascular Closure System
Other: Manual Compression — manual pressure applied to your groin for approximately 5-10 minutes
  Arms: Manual Compression

SUMMARY:
Evaluate the safety of the MynxGrip™ extravascular sealant for common femoral vein closure following both diagnostic and interventional procedures as assessed by clinical and imaging criteria.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety of the MynxGrip™ extravascular sealant for common femoral vein closure following both diagnostic and interventional procedures as assessed by clinical and imaging criteria for venous thrombosis at the site of closure device deployment.

This is a single-center prospective study of patients who are undergoing either diagnostic or interventional procedures. A total of 208 patients will be enrolled in this study and will be followed through hospital discharge for safety purposes.

The primary safety endpoint will include both deep venous thrombotic and bleeding/vascular injury related complications prior to discharge. Outcomes will be assessed via clinical evaluation and imaging with clinically indicated as follow:

Assessment of venous thrombosis i. Clinical: Physical exam findings consistent with venous thrombotic/thromboembolic related complication:

* Redness or swelling at the venous puncture site
* Increased lower extremity edema
* Calf pain
* New onset or worsening shortness of breath
* New onset of pleuritic chest pain ii. and if clinically indicated, imaging: venous Doppler ultrasound assessment of obstructive or non-obstructive deep vein thrombosis (DVT)

  * Bleeding or vascular related complications i. Damage to the vessel requiring surgical repair ii. Access site bleeding requiring the need for transfusion iii. Nerve injury at access site iv. Generalized infection (septicemia with typical signs, symptoms and positive blood cultures shortly after the index procedure, and requiring treatment with intravenous (IV) antibiotics)Pseudo-aneurysms requiring invasive treatment
  * Device/procedure failure Device failure is defined as either the inability to deploy the device or device deployment with inadequate hemostasis requiring conversion to immediate manual pressure, or the eventual need for alternative methods to obtain hemostasis.

Efficacy will be assessed by time to hemostasis; Time to hemostasis is defined as the time from advancer tube removal (i.e., device removal) to the time when hemostasis was first observed.

The study will be conducted following either diagnostic or interventional procedures where venous access was required (via the common femoral vein with insertion of 5, 6, or 7F sheath). Femoral vein hemostasis will be achieved with either manual compression or the MynxGrip VCD system. To assess the primary safety outcome of venous patency and lack of occurrence of DVT, clinical assessment will be performed by the study team vascular access assessment group and when clinically indicated a duplex ultrasound will be performed on patients prior to discharge to evaluation the presence of venous thrombosis.

After enrollment, subjects will be randomized 1:1 to:

* Treatment Group A: Subjects will have venous hemostasis achieved using the MynxGrip vascular closure system in the common femoral vein.
* Treatment Group B: Subjects will have venous hemostasis achieved using manual compression over the common femoral vein.

Subjects who meet all inclusion criteria and none of the exclusion criteria, who agree to participate in this clinical study, and who sign an informed consent will be enrolled.

The patient will undergo the clinically indicated procedure(s) as per standard of care. The type of procedure(s) performed will be collected within the CRF. Once all the clinically indicated procedures have been completed the following assessment will be made with respect to the inclusion criteria:

* Target vein had a maximal sheath size inserted larger that 7Fr
* Multiple (>1) attempts at venous access were attempted in the target vein
* Patient has intra-procedural bleeding around the access site prior to sheath removal
* Critically ill patients requiring intravenous vasopressors for blood pressure stabilization
* Ipsilateral femoral artery puncture or sheath insertion
* Glycoprotein IIb/IIIIa use
* Any bleeding or vascular access-site complication evident pre-venous closure If any of the above are met, then the patient will be considered a screen failure. If one femoral vein was attempted with one or more access attempts with or without sheath insertion and then the contralateral femoral vein is used to gain venous access, the target vein for closure would become the vein with one attempt to achieve access that also fits the inclusion/ exclusion criteria above.

Randomization and Enrollment Once the patient meets all the inclusion criteria and none of the exclusion criteria he/she will be considered enrolled in the study.

Randomization will be performed in a block size of 4 within site to maintain the 1:1 randomization throughout the trial within two patients. Randomization will be assigned in consecutive order for the patient enrollment ID starting with 001 through 208. The randomization assignment will be stored within an opaque envelope and assigned/opened in numerical order.

Study Devices/ Procedures

For the randomization assignments both commercial product will be uses. Please follow the commercial IFU for deployment and/or positioning of the Mynx Vascular Closure. For manual compression please follow the local institutions standard of care for the procedure.

Follow-up Patients will be followed up though hospital discharge to assess the primary safety outcome of deep vein thrombotic and/or bleeding/vascular injury related complications related to the target venous closure site.

To assess this primary safety outcome of venous patency and lack of occurrence of DVT, a clinical assessment this includes the following by systematic physician assessment of the target groin.

Once the patient is placed in the recovery room following the completion of the procedure, a member of the Mynx Grip study team will be called to assess the groin, which includes the information below;

Assessment of Venous Thrombosis:

* Comparing mid calf and mid thigh measurement prior to and post procedure.
* Redness or selling at the venous puncture site
* Physical exam findings consistent with venous thrombotic/thromboembolic related complications (i.e. vein engorgement, presence of chord, syenosis)
* Increased lower extremity edema
* New onset or worsening shortness of breath
* New onset of pleuritic chest pain

Bleeding or Vascular Related complications:

* Damage to the vessel requiring surgical repair
* Access site bleeding requiring the need for transfusion
* Nerve injury at the access site
* Generalized infection
* Pseudo-aneurysms requiring invasive treatment In the event that the Mynx Grip study team believes that further assessment for venous thrombosis of the target femoral vein is necessary, a duplex ultrasound of the target femoral vein will be ordered.

Presence of a venous thrombosis of the target vein will be assessed based on a combination of clinical symptoms and/or result of the duplex ultrasounds. Duplex ultrasounds will be submitted to and assessed by the Duplex Ultrasound Core Lab for a systematic and objective review of the presence of venous thrombosis

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age scheduled for a percutaneous diagnostic or interventional procedure that have either a 5, 6, or 7F sheath placed in the common femoral vein.

Exclusion Criteria:

1. Patient has a history of a bleeding disorder
2. Previous history of venous thrombosis or thromboembolism
3. Patient is pregnant or lactating
4. Patient has a known severe allergy to contrast medium
5. Patient has a known allergy to PEG

7. Patient is known to require an extended hospitalization or re-hospitalization (e.g. patient is undergoing coronary artery bypass graft (CABG) surgery) or patient is scheduled to have a CABG surgery <30 days following the procedure) 9. Multiple (>1) attempts at venous access were attempted in the target vein 10. Patient has intra-procedural bleeding around the access site prior to sheath removal 11. Critically ill patients requiring intravenous vasopressors for blood pressure stabilization 12. Ipsilateral femoral artery puncture or sheath insertion 13. Glycoprotein IIb/IIIIa use 14. Any bleeding or vascular access-site complication evident pre-venous closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2015-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Southern Maryland Hospital, Clinton, Maryland

REFERENCES:
- [Result] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Result] Tavris DR, Dey S, Albrecht-Gallauresi B, Brindis RG, Shaw R, Weintraub W, Mitchel K. Risk of local adverse events following cardiac catheterization by hemostasis device use - phase II. J Invasive Cardiol. 2005 Dec;17(12):644-50. PMID 16327045
- [Result] Marso SP, Amin AP, House JA, Kennedy KF, Spertus JA, Rao SV, Cohen DJ, Messenger JC, Rumsfeld JS; National Cardiovascular Data Registry. Association between use of bleeding avoidance strategies and risk of periprocedural bleeding among patients undergoing percutaneous coronary intervention. JAMA. 2010 Jun 2;303(21):2156-64. doi: 10.1001/jama.2010.708. PMID 20516416
- [Result] Scheinert D, Sievert H, Turco MA, Schmidt A, Hauptmann KE, Mueller R, Dadourian D, Krankenberg H, Grube E. The safety and efficacy of an extravascular, water-soluble sealant for vascular closure: initial clinical results for Mynx. Catheter Cardiovasc Interv. 2007 Nov 1;70(5):627-33. doi: 10.1002/ccd.21353. PMID 17960627
- [Result] Zahn R, Fromm E, Thoma S, Lotter R, Zander M, Wagner S, Seidl K, Senges J. Local venous thrombosis after cardiac catheterization. Angiology. 1997 Jan;48(1):1-7. doi: 10.1177/000331979704800101. PMID 8995337

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mynx Vascular Closure System | Manual Compression
Started | 104 | 104
Completed | 102 | 104
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mynx Vascular Closure System | Manual Compression | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 26 | 48
  >=65 years | 82 | 78 | 160
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 91
  Male | 61 | 56 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 32 | 52
  White | 83 | 69 | 152
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 104 | 104 | 208

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Venous Thrombosis
Description: i. Clinical: Physical exam findings consistent with venous thrombotic/thromboembolic related complication:
  * Redness or swelling at the venous puncture site
  * Increased lower extremity edema
  * Calf pain
  * New onset or worsening shortness of breath
  * New onset of pleuritic chest pain ii. and if clinically indicated, imaging: venous Doppler ultrasound assessment of obstructive or non-obstructive deep vein thrombosis (DVT)
Time Frame: Subjects will be followed up until their discharge from the hospital, and expected average of 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Mynx Vascular Closure System | Manual Compression
Number analyzed (Participants) | 103 | 104
Participants | 0 | 0

2. Primary Outcome: Bleeding or Vascular Related Complications
Description: i. Damage to the vessel requiring surgical repair ii. Access site bleeding requiring the need for transfusion iii. Nerve injury at access site iv. Generalized infection (septicemia with typical signs, symptoms and positive blood cultures shortly after the index procedure, and requiring treatment with intravenous (IV) antibiotics)Pseudo-aneurysms requiring invasive treatment
Time Frame: Subjects will be followed up until their discharge from the hospital, and expected average of 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Mynx Vascular Closure System | Manual Compression
Number analyzed (Participants) | 103 | 104
Participants | 0 | 0

3. Primary Outcome: Device/Procedure Failure
Description: Device failure is defined as either the inability to deploy the device or device deployment with inadequate hemostasis requiring conversion to immediate manual pressure, or the eventual need for alternative methods to obtain hemostasis.
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Mynx Vascular Closure System | Manual Compression
Number analyzed (Participants) | 103 | 104
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: procedure through hospital discharge
Arm/Group | Mynx Vascular Closure System | Manual Compression
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 7/104 | 15/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mynx Vascular Closure System (N=104) | Manual Compression (N=104)
Access site thigh change >2 cm (Blood and lymphatic system disorders) | 7 (7) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02438475/Prot_SAP_000.pdf